CLINICAL TRIAL: NCT07194577
Title: "Effect of Moringa Oleifera Dehydrated Leaf Powder on the Components of Metabolic Syndrome in Mexican Adults. Double-blind Randomized Clinical Trial. Phase II"
Brief Title: Effect of Moringa Oleifera Dehydrated Leaf Powder on the Components of Metabolic Syndrome in Mexican Adults.
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Colima (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CarmenSanchez, Principal Investigator, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOD
Record Dates: First submitted 2025-05-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Nutritional and Metabolic Diseases; Metabolic Syndrome
Keywords: Metabolic syndrome; Moringa oleifera; Diabetes Mellitus type 2; Dyslipidemia
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Metabolic Syndrome; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Intervention Model Description: 42 adults diagnosed with metabolic syndrome will be randomly assigned to either the intervention group or the placebo group. The data collected will be weight, height, blood pressure, and waist circumference, and blood tests include glucose, lipid profile [triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol], and glycosylated hemoglobin. Both groups will be evaluated before starting treatment and 8 weeks later, after completing the treatment.
Who Masked: Participant, Investigator
Masking Description: Computer-generated random numbers will be used for simple randomization of subjects to the intervention group and placebo group, which will be performed by someone unrelated to the investigation and provided to the principal investigator in closed envelopes with 2 different categories (A or B), so that the principal investigator does not know the group to which the study subjects belong. Likewise, patients will recieve their treatment marked as A or B, but will not know which group they belong to (experimental or placebo) until the final results of the study are available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moringa oleifera (Experimental): To determine if Moringa oleifera dried leaf powder has an effect * in the components of metabolic syndrome in adults compared to placebo.
  5.5 grams of Moringa oleifera Lam leaf powder per day (9 capsules with 0.6 g each) divided into 3 doses - 3 with breakfast, 3 with lunch, 3 with dinner - daily for 8 weeks.
  Interventions: Dietary Supplement: Moringa oleifera
- Placebo (Placebo Comparator): To determine if Moringa oleifera dried leaf powder has an effect * in the components of metabolic syndrome in adults compared to placebo.
  Starch capsules, (9 capsules with 0.6 g each) divided into 3 doses - 3 with breakfast, 3 with lunch, 3 with dinner - daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Moringa oleifera — 5.6 grams of Moringa oleifera Lam dried leaf powder administered orally per day (as nine 0.5 g capsules), divided into three doses (three capsules with breakfast, three with lunch, and three with dinner) for 8 weeks.
  Arms: Moringa oleifera
Dietary Supplement: Placebo — Starch placebo administered orally per day (as nine 0.5 g capsules), divided into three doses (three capsules with breakfast, three with lunch, and three with dinner) for 8 weeks.
  Arms: Placebo

SUMMARY:
Background: The increase in chronic degenerative diseases caused by Metabolic Syndrome (MS) has prompted the search for natural alternatives to develop new medications and to know the mechanism and dosages for their proper use. To date, evidence of the potential use of moringa in the context of metabolic diseases such as diabetes mellitus 2, obesity, and dyslipidemia is available. However, before they can be used as a treatment for metabolic diseases in humans, clinical studies must be carried out to establish the consistency of its medicinal efficacy and the safest modalities of its administration. Objective: To compare the effect of Moringa oleifera dehydrated leaf powder vs a placebo on the components of metabolic syndrome in mexican adults. Material and methods: Double blind randomized clinical trial, phase II. 42 adults diagnosed with MS treated at the family medical consultation of Clinic 19 of the IMSS Colima will be randomly assigned to 2 groups: intervention group (MO powdered leaf capsules, 5.5 grams per day) and placebo group (starch capsules, 5.5 grams per day). The data collected will be weight, height, blood pressure, and waist circumference, and blood tests include glucose, lipid profile [triglycerides, total cholesterol, HDL cholesterol], glycosylated hemoglobin. Both groups will be evaluated before starting treatment and 8 weeks later, after completing the treatment. Resources and infrastructure: The laboratory exams will are carried out in HGZ1 no.1 of the IMSS.

DETAILED DESCRIPTION:
1. . Data collection. The patients are being recruited from the medical consultation of the UMF 19 of the IMSS Colima. Participants must have a previous Metabolic Syndrome diagnosis in their medical record (3 or more diagnostic variables according to the 2009 standarization by the International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity).
2. . Study groups. 1) Intervention group [moringa oleifera leaf powder capsules of 0.6 g each]. 5.5 grams a day divided into 3 doses: 3 capsules of 0.6 g each in the morning, 3 capsules of 0.6 g each in the afternoon, 3 capsules of 0.6 g each at night]. 2) Placebo group [5.5 grams of placebo (corn starch) per day divided into 3 doses: 3 capsules of 0.6 g each in the morning, 3 capsules of 0.6 g each in the afternoon, 3 capsules of 0.6 g each at night].
3. . Randomization and blinding. Computer-generated random numbers were used for simple randomization of subjects to the intervention group (Group A) and placebo group (Group B). Neither the patients nor the principal investigator know to which group subjects belong to (experimental or placebo) until the final results of the study are available.
4. . Preparation of treatment and placebo. For the present study, a sample size of 42 patients was calculated. Each person will consume nine capsules #00 per day (0.63 g each) for a period of 8 weeks. 504 capsules per person will be needed, which is equivalent to a total of 21,168 capsules , of which 10,584 will be Moringa oleifera leaf powder and 10,584 corn starch as an excipient. Due to the nature of the study (double blind), all capsules are black so there is no way to see the contents inside the capsules. Both the raw material (#00 capsules, Moringa oleifera leaf powder (10 kg), starch (10 kg)) and the encapsulation service were provided by the company Encapsuladoras México, based in Chihuahua, Chihuahua. This guarantees a quality product with excellent hygiene standards and precision in the content of the capsules.
5. . Follow-up and adherence to treatment. Both groups (A and B) undergo baseline analyzes before receiving any treatment to ensure that they meet the inclusion criteria and have no metabolic or organ risk. In case of corroborating any lack of control in a patient (monitored with the baseline analysis), the treating physician will make the pertinent adjustment with the medications according to the guidelines and procedures of the HGZ No. 1 of the IMSS Colima. Both groups receive their total capsule doses (504 capsules) divided into two doses with 252 capsules each (one dose for each month). The daily dose contain 5.5 g of Moringa oleifera or placebo (corn starch). Participants are instructed to consume 9 capsules per day divided into 3 doses: 3 capsules in the morning, 3 capsules in the afternoon, 3 capsules in the evening; capsules should be taken before each corresponding meal time (breakfast, lunch, dinner). This goes on for a period of 8 weeks. The delivery of the capsules takes place outside the medical consultation of the Family Medical Unit #19 of the IMSS Colima once the results of the baseline laboratory analyzes are obtained. First month of treatment is given, the patients are summoned again and the following month of treatment is given. To ensure a minimum adherence of 80%, a weekly format is given to the participants together with the capsules. Fort he follow-up, a Whatsapp group was created for motivation and weekly reminders, and phone calls are made once a week to answer questions and find out about follow-up. At the end of their treatment, the participants are summoned again to take final measurements and laboratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries of the medical consultation of the Instituto Mexicano del Seguro Social (IMSS), Colima
* - Female and male gender
* People with 3 diagnostic variables of metabolic syndrome according to the standardization of criteria established for the diagnosis of Metabolic Syndrome (2009).
* Patients under treatment for components of metabolic syndrome (dyslipidemia, diabetes, arterial hypertension)
* Signed informed consent

Exclusion Criteria:

* Conditions that do not allow blood collection
* Patients with metabolic syndrome who currently follow a nutritional plan and/or do exercise
* Pregnant women
* Smokers
* Patients with hypothyroidism and hyperthyroidism, cancer, renal failure and/or liver cirrhosis
* Patients with any complication of diabetes mellitus
* Patients on insulin therapy
* People who take botanical extracts or a multivitamin
* People with food allergies
* Acute infection in progress at the time of blood sample collection
* Patients must not be participating in another study alternately

Elimination Criteria

* Insufficient, coagulated or hemolyzed serum sample.
* Patients who interrupt treatment or who do not wish to continue.
* Patients who present side effects (nausea, vomiting, diarrhea, stomach pain) or any symptom related to discomfort, allergy or intolerance with the consumption of Moringa oleifera leaf powder that does not disappear in a period of 3 days.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the prevalence of Metabolic Syndrome | 8 weeks
  The change in the proportion of participants meeting the diagnostic criteria for Metabolic Syndrome (according to the NCEP ATP III citeria) from baseline to 8 weeks. The outcome is reported as the difference in prevalence rates between the intervention and placebo groups.

SECONDARY OUTCOMES:
Compare the effect of body mass index (BMI) in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention endsThis measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2.
  BMI classification kg/m2:
  Normal range 18.5-24.9 Overweight > 25 Obesity > 30 (82). According to the WHO (2023) and the NIH (2022), an absolute reduction of ≥5% from the initial BMI is considered clinically relevant in the general population, ≥10% in people with obesity (BMI ≥30) or comorbidities (diabetes, hypertension) A reduction of ≥5% between the baseline and final measurements will be considered an improvement.
Compare the effect of waist circumference in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Waist circumference for Hispanics >94 cm in men and >88 cm in women. A 5-10% reduction from baseline WC improves insulin sensitivity and lipid profile. The formula is calculated as follows:
  Percentage reduction = [(baseline value - final value)/ baseline value] x 100
Compare the effect of blood pressure in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Elevated systolic blood pressure values is >130 mmHg, and is associated with an increased risk of organ damage and cardiovascular events. A reduction in SBP >5 mmHg between baseline and final measurement will be considered an improvement.
  Elevated diastolic blood pressure is >85 mm/Hg (Antihypertensive drug treatment in a patient with a history of hypertension is an alternative indicator). A reduction in DAS >3 mm/Hg between baseline and final measurement will be considered improvement.
Compare the effect of fasting glucose in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Elevated fasting glucose >100 mg/dL (Pharmacological treatment for elevated glucose is an alternative indicator). The American Diabetes Association (ADA) and the World Health Organization (WHO) consider a clinically significant improvement in studies with natural interventions (such as Moringa oleifera) when there is a reduction in fasting glucose of ≥20 mg/dL (1.1 mmol/L) in the diabetic population, or ≥10 mg/dL (0.55 mmol/L) in prediabetes.
  A reduction of ≥10 mg/dL between the baseline and final measurement will be considered an improvement.
Compare the effect of HDL-Cholesterol in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Adequate values for men: <40 mg/dL (1.0 mmol/L); for women: <50 mg/dL (1.3 mmol/L) (Pharmacological treatment for reduced HDL-C is an alternative indicator). According to the AHA/ACC and NLA guidelines (2023), a clinically relevant improvement is considered to be an absolute increase in HDL of ≥5 mg/dL (0.13 mmol/L) in the general population, and ≥10 mg/dL (0.26 mmol/L) in patients with diabetes or metabolic syndrome.
  An increase of ≥5 mg/dL between the baseline and final measurements will be considered an improvement.
Compare the effect of triglycerides in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Normal values >150 mg/dL (1.7 mmol/L) (Pharmacological treatment for elevated triglycerides is an alternative indicator). According to the AHA/ACC (2023) and the National Lipid Association (2023), a 20-30% percentage reduction is considered clinically relevant. The formula is calculated as follows:
  Percent reduction = [(baseline value - final value)/ baseline value] x 100
Compare the effect of total cholesterol in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Normal values <200 mg/dL Reduction will be considered of 5-10% from baseline. The formula used is Percent reduction = [(baseline value - final value)/ baseline value] x 100
  baseline value
Compare the effect of LDL-Cholesterol in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Normal values <100 mg/dL.
  Change is 30-50% reduction from baseline (for statins or combination therapies) . The formula is calculated as follows:
  Percent reduction = [(baseline value - final value) / baseline values] x 100
Compare the effect of non- HDL-Cholesterol in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  Normal values <130 mg/dL .
  Change is 20-30% reduction from baseline. The formula is calculated as follows:
  Percent reduction = [(baseline value - final value)/ baseline value] x 100
Compare the effect of glycated hemoglobin in the experimental group vs. placebo group | This measurement will be taken at the beginning of the protocol, and then 8 weeks later, when the intervention ends
  According to the American Diabetes Association, a diagnosis of type 2 diabetes based on glycated hemoglobin is made when HbA1c is 6.5% or higher, and high risk of this condition is present with an HbA1c of 5.7-6.4%. A reduction in HbA1c of >0.5% between baseline and final measurement is considered an improvement in diabetic patients.
  A reduction of ≥0.5% between baseline and final measurement will be considered an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Iván Delgado Enciso, Doctor, Study Director — Universidad de Colima; Carmen Alicia Sánchez Ramírez, Doctor, Study Director — Universidad de Colima
Locations (1):
- Unidad de Medicina Familiar No.19, Instituto Mexicano del Seguro Social, Colima, Centro, Mexico

IPD SHARING:
Plan to Share IPD: No
At the moment we will not share the information until having preliminary results.

REFERENCES:
- [Background] Writing Committee Members; Virani SS, Newby LK, Arnold SV, Bittner V, Brewer LC, Demeter SH, Dixon DL, Fearon WF, Hess B, Johnson HM, Kazi DS, Kolte D, Kumbhani DJ, LoFaso J, Mahtta D, Mark DB, Minissian M, Navar AM, Patel AR, Piano MR, Rodriguez F, Talbot AW, Taqueti VR, Thomas RJ, van Diepen S, Wiggins B, Williams MS. 2023 AHA/ACC/ACCP/ASPC/NLA/PCNA Guideline for the Management of Patients With Chronic Coronary Disease: A Report of the American Heart Association/American College of Cardiology Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2023 Aug 29;82(9):833-955. doi: 10.1016/j.jacc.2023.04.003. Epub 2023 Jul 20. PMID 37480922
- [Background] Taweerutchana R, Lumlerdkij N, Vannasaeng S, Akarasereenont P, Sriwijitkamol A. Effect of Moringa oleifera Leaf Capsules on Glycemic Control in Therapy-Naive Type 2 Diabetes Patients: A Randomized Placebo Controlled Study. Evid Based Complement Alternat Med. 2017;2017:6581390. doi: 10.1155/2017/6581390. Epub 2017 Nov 28. PMID 29317895
- [Background] Haber SL, McMahon RP, Barajas J, Hayes AR, Hussein H. Effects of Moringa oleifera in patients with type 2 diabetes. Am J Health Syst Pharm. 2020 Oct 30;77(22):1834-1837. doi: 10.1093/ajhp/zxaa255. No abstract available. PMID 32960218
- [Background] Chan Sun M, Ruhomally ZB, Boojhawon R, Neergheen-Bhujun VS. Consumption of Moringa oleifera Lam Leaves Lowers Postprandial Blood Pressure. J Am Coll Nutr. 2020 Jan;39(1):54-62. doi: 10.1080/07315724.2019.1608602. Epub 2019 May 7. PMID 31063434
- [Background] Wang F, Bao Y, Zhang C, Zhan L, Khan W, Siddiqua S, Ahmad S, Capanoglu E, Skalicka-Wozniak K, Zou L, Simal-Gandara J, Cao H, Weng Z, Shen X, Xiao J. Bioactive components and anti-diabetic properties of Moringa oleifera Lam. Crit Rev Food Sci Nutr. 2022;62(14):3873-3897. doi: 10.1080/10408398.2020.1870099. Epub 2021 Jan 6. PMID 33401950
- [Background] Gomez-Martinez S, Diaz-Prieto LE, Vicente Castro I, Jurado C, Iturmendi N, Martin-Ridaura MC, Calle N, Duenas M, Picon MJ, Marcos A, Nova E. Moringa oleifera Leaf Supplementation as a Glycemic Control Strategy in Subjects with Prediabetes. Nutrients. 2021 Dec 24;14(1):57. doi: 10.3390/nu14010057. PMID 35010932
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- See also: International Diabetes Federation. (2023). IDF Consensus Worldwide Definition of the Metabolic Syndrome. — https://www.idf.org
- See also: World Health Organization. (2023). Obesity and overweight. — https://www.who.int